CLINICAL TRIAL: NCT05503212
Title: Best Revascularisation Approach for Posterior Circulation Strokes With Isolated Vertebral : the BRAVO Retrospective Analysis
Brief Title: Best Revascularisation Approach for Posterior Circulation Strokes With Isolated Vertebral Artery Occlusions
Acronym: BRAVO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Asan Medical Center (Other); St John of God Hospital, Vienna (Other); Medical University Innsbruck (Other); Hospital Vall d'Hebron (Other); University Hospital, Basel, Switzerland (Other); Clinical Centre of Serbia (Other); Charite University, Berlin, Germany (Other); Insel Gruppe AG, University Hospital Bern (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Boston Medical Center (Other); Università degli Studi di Brescia (Other); The Cooper Health System (Other); University Hospital Carl Gustav Carus (Other); Duke University (Other); University Hospital, Geneva (Other); Hadassah Medical Organization (Other); Sahlgrenska University Hospital (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Helsinki University Central Hospital (Other); The University of Texas Health Science Center, Houston (Other); University Hospital, Lille (Other); Hospital de Egas Moniz (Other); Neurocenter of Southern Switzerland (Other); Corewell Health West (Other); Azienda Ospedaliero-Universitaria di Modena (Other); Ludwig-Maximilians - University of Munich (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); University of Zurich (Other)
Responsible Party: Principal Investigator, Dr. med. Alexander Salerno, MD, Clinical Researcher, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: Stroke-VAO
Record Dates: First submitted 2022-03-22; First posted 2022-08-16 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Ischemic Stroke; Vertebral Artery Ischemia; Arterial Occlusive Diseases; Vertebrobasilar Insufficiency
Keywords: Prognosis; Revascularization; Treatment
MeSH Terms: conditions — Ischemic Stroke; Vertebrobasilar Insufficiency; Arterial Occlusive Diseases | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AIS and isolated VAO: Patients with acute ischemic stroke (AIS) and concomitant isolated intracranial and/or extracranial vertebral artery occlusion (VAO)
  Interventions: Other: Conservative treatment (CT); Other: Intravenous thrombolysis (IVT); Other: Endovascular thrombectomy (EVT) ± intravenous thrombolysis (IVT)

INTERVENTIONS:
Other: Conservative treatment (CT) — Best medical treatment without intravenous thrombolysis nor endovascular thrombectomy
Other: Intravenous thrombolysis (IVT) — Best medical treatment with intravenous thrombolysis but without endovascular thrombectomy
Other: Endovascular thrombectomy (EVT) ± intravenous thrombolysis (IVT) — Best medical treatment with endovascular thrombectomy with or without intravenous thrombolysis

SUMMARY:
Isolated vertebral artery occlusions (VAO) account for approximately one third of posterior circulation occlusions, but have been given the least attention among posterior circulation strokes. If the two recent ATTENTION and BAOCHE randomized clinical trials have proven the superiority of endovascular thrombectomy (EVT) in basilar artery occlusions, data on the effectiveness and harm of acute revascularization treatment on isolated VAO is scarce. We aim to investigate the impact of acute recanalisation treatments in acute ischemic stroke patients with isolated VAO.

In the absence of RCT, observational data with appropriate statistical methods may give indications on benefits and harms of treating neglected stroke situations like acute vertebral occlusion. Results may also lay the basis for prospective studies, such as randomized clinical trials.

ELIGIBILITY:
Inclusion criteria:

* Acute ischemic stroke limited to the posterior circulation
* Presence of uni- or bilateral VAO (intracranial and/or extracranial) on at least one initial imaging study (CTA, MRA, DSA)
* IVT, EVT or bridging-treated stroke patients between 01.01.2003 and 31.12.2021
* ≥ 18 years old

Exclusion criteria

* Extension of the occlusion into the basilar artery
* Presence of a more distal occlusion in the pc (tandem occlusion/multilevel poster circulation occlusions)
* Previously known chronic occlusion of the any segment of the vertebral artery/arteries
* Local ethical/legal conditions in participating center not fulfilled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke and concomitant isolated vertebral artery occlusion accounting for stroke symptoms
Sampling Method: Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
3-month modified Rankin scale | 90 days
  3-month functional outcome, [range: 0-6, 0= no symptoms, 6=death]

SECONDARY OUTCOMES:
Symptomatic intracerebral haemorrhage (sICH) | 7 days
  Any hemorrhagic transformation temporally related to any worsening in neurological condition. [yes/no]
EVT procedural complications | During EVT procedure or peri-procedural
  Any complication attributed to the procedure (vessel perforation, vasospasm, dissection, Subarachnoid haemorrhage (SAH)/Intracerebral haemorrhage (ICH), device detachment/misplacement, embolization to new territory, access-site complications, early reocclusion, other)
24-hour NIHSS | 24 hours
  NIH Stroke Scale/Score (NIHSS). Quantifies stroke severity based on weighted clinical evaluation findings at 24h. [0-42, 0= no deficit, 42=maximum stroke severity]
Early neurological deterioration (ENDi) | 24 hours
  Early neurological deterioration of ischemic origin (ENDi) is defined as an increase in National Institute of Health Stroke (NIHSS) score ≥ 4 points or death within 24 hours. [yes/no]
Cerebrovascular ischemic recurrences | 90 days
  Any ischemic stroke or transient ischemic attack recurrence [yes/no]
24h and 3month mortality | 24h and 90 days
  Mortality at 24h and 3 months
Vessel recanalisation on follow up-imaging | 48 hours
  Vessel recanalisation at follow-up imaging (0= no recanalisation, 1= partial recanalisation 50-99%, 2=full recanalisation, 3= initially not occluded)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med. Alexander Salerno, MD, Principal Investigator — CHUV
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland